CLINICAL TRIAL: NCT05362305
Title: Essential Coaching for Every Mother: Developing and Evaluating a Text Message Postnatal Education Intervention for Mothers of Newborns in Tanzania
Brief Title: Essential Coaching for Every Mother in Tanzania
Acronym: ECEMTZ
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Principal Investigator, Justine Dol, Principal Investigator, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ECEMTZ
Record Dates: First submitted 2022-04-22; First posted 2022-05-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Parenting Self Efficacy; Postpartum Depression; Postpartum Anxiety; Breastfeeding Self-Efficacy; Newborn Knowledge
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Essential Coaching for Every Mother (Experimental): Mothers in the intervention group will receive in-hospital education by a non-study nurse midwife while on the postnatal ward prior to discharge as per standard protocol on the unit. On the third day after birth, mothers will receive daily text messages to 6 weeks postpartum. The messages will be sent automatically each day based on the date of birth of the infant.
  Interventions: Behavioral: Essential Coaching for Every Mother
- Standard Care (No Intervention): Mothers will receive in-person education provided by a non-study nurse midwife while on the postnatal ward prior to discharge as per current standard protocol on the unit. Mothers in this group will not receive any further text messages from the program.

INTERVENTIONS:
Behavioral: Essential Coaching for Every Mother — Daily text messages for the first six-weeks postpartum.
  Arms: Essential Coaching for Every Mother

SUMMARY:
The purpose of this study is to evaluate a text message intervention called Essential Coaching for Every Mother in Tanzania to improve mothers' access to essential newborn care information during the immediate six-week postnatal period.

DETAILED DESCRIPTION:
This is a 2-group parallel arm randomized controlled trial. Participants will be randomized into either the intervention or a control group. No changes to in-person care will occur.

This study will be conducted in Dar es Salaam, Tanzania with mothers recruited from a Tanzanian postnatal ward who have recently given birth at four different hospitals. Participants in the intervention group will start receiving the Essential Coaching for Every Mother program based on their delivery date up to six weeks postpartum. Mothers in the control group will not receive any text messages. Both groups will be asked to complete a survey at enrolment and six-weeks postpartum.

The investigators aim to recruitment 124 participants in total, 62 per group.

ELIGIBILITY:
Inclusion Criteria:

* have recently given birth within the hospital within 48 hours
* have daily access to a mobile phone with text message capabilities
* are over 18 years of age
* speak and read English or Swahili.

Exclusion Criteria:

* newborns die or are expected to die prior to leaving the hospital
* they have no access to mobile phone, either personal or shared
* unwilling to receive text messages
* decline to participate
* are experiencing major postnatal complications expected to impact learning or ability to consent while in the hospital (e.g., postpartum hemorrhage, seizures)
* participated in Phase I of this project.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2024-09-21 (Actual); Study Completion 2025-10-10 (Estimated)

PRIMARY OUTCOMES:
Newborn Care Knowledge | Baseline (enrolment), and six-weeks postpartum (follow-up)
  Knowledge will be assessed using a modified questionnaire developed by McConnell and colleagues. Questions will determine whether mothers can identify danger signs, hand washing practices, cord care, newborn thermal care, and breastfeeding. A summative score will be created with a maximum of five points and a minimum of zero, where each point represents knowledge on the above postnatal health topics.

SECONDARY OUTCOMES:
Maternal Self-Efficacy | Baseline (enrolment), and six-weeks postpartum (follow-up)
  Parenting self-efficacy will be measured using the Karitane Parenting Confidence Scale (KPCS) tool. This 15-item tool was developed to assess perceived self-efficacy of mothers of newborns birth to twelve months of age. A cut off score of 39 or less (out of a possible 45) was determine to be a clinically low perceived parenting self-efficacy (PPSE).
Breastfeeding Self-Efficacy | Baseline (enrolment), and six-weeks postpartum (follow-up)
  Breastfeeding self-efficacy will be measured using the Breastfeeding Self-Efficacy Scale - Short Form. Higher scores indicate higher breastfeeding self-efficacy.
Postpartum Depression | Baseline (enrolment), and six-weeks postpartum (follow-up)
  Depression will be measured using the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a self-report screening scale with 10 items that can indicate if a respondent has symptoms related to perinatal depression with a score >12 considered high symptoms of depression.
Postpartum Anxiety | Baseline (enrolment), and six-weeks postpartum (follow-up)
  Anxiety will be measured using the Generalized Anxiety Disorder (GAD)-7, which is a 7-item scale used to assess generalized anxiety disorder. The scale ranges between 0 and 21, with scores of 10 or greater indicative of generalized anxiety at a moderate/severe level.
Newborn morbidity | Six-weeks postpartum (follow-up)
  Data will be collected on number of morbidities (e.g., diarrhea, jaundice, infection) identified per infant enrolled in the study within the 6-weeks.
Newborn mortality | Six-weeks postpartum (follow-up)
  Data will be collected on newborn mortality (e.g., number of infant deaths during study).
Need for readmission | Six-weeks postpartum (follow-up)
  Data will be collected on number of readmission to hospital for the infant and mothers during the six weeks and related reason.
Postnatal Clinic Attendance | Six-weeks postpartum (follow-up)
  Data will be collected on the number and date of postnatal contact.

OTHER OUTCOMES:
Implementation Dose | Enrolment and study completion (6 weeks)
  Dose delivered - number of text messages sent. Output data available through the Africa's Talking and TextIt platforms will be collected per participant.
Implementation Engagement | Enrolment and study completion (6 weeks)
  Un-subscription rates/drop out after enrolment. Output data available through the Africa's Talking and TextIt platforms will be collected per participant.
Recruitment Effectiveness | Enrolment
  Number of participants enrolled versus approached. Number of participants per hospital site.
Implementation Quality | Six-weeks postpartum
  Mothers in the intervention group will be asked about the number of messages they recall receiving, user experience, perspectives on the frequency and timing of messages, and what did they like and not like about Essential Coaching for Every Mother.

CONTACTS AND LOCATIONS:
Locations (1):
- Muhimbili University of Health and Allied Sciences, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dol J, Mselle LT, Campbell-Yeo M, Mbekenga C, Kohi T, McMillan D, Dennis CL, Tomblin Murphy G, Aston M. Essential Coaching for Every Mother Tanzania (ECEM-TZ): Protocol for a Type 1 Hybrid Effectiveness-Implementation Randomized Controlled Trial. JMIR Res Protoc. 2024 Dec 5;13:e63454. doi: 10.2196/63454. PMID 39636672